CLINICAL TRIAL: NCT04042363
Title: Effect of Transorbital Electrical STIMulation of Optic Nerve on Remyelination After an Acute Optic Neuritis
Acronym: ONSTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Collaborators: Fondation ARSEP (Unknown); APHP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P18-03; 2018-A03138-47 (Other: ID RCB)
Record Dates: First submitted 2019-07-16; First posted 2019-08-01 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis; Optic Neuritis
Keywords: multiple sclerosis; optic neuritis; transorbital stimulation; remyelination; nervous system disease; peripheral nervous system disease; optic nerve disease; adaptive optic
MeSH Terms: conditions — Multiple Sclerosis; Optic Neuritis; Nervous System Diseases; Peripheral Nervous System Diseases; Optic Nerve Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients as well as ophthalmologists will be subject to the procedure of masking and will keep the blinding for the duration of the study. As a result, ophthalmologists examiners will not perform electrical stimulation sessions.
  The persons in charge of the stimulation will be in "open label" and will ensure the inclusion, the follow-up of the patient throughout the study, the stimulation (SHAM or stimulation), the clinical and neurological examination as well as the collection of the treatments and the notification of the Adverse Events/Serious Adverse Events (AE/SAE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transorbital electrical stimulation (Experimental): Transorbital electrical stimulation of the optic nerve - 10 sessions during 2 consecutive weeks
  Interventions: Device: Transorbital electrical stimulation (Eyetronic Next Wave 1.1)
- Sham Transorbital stimulation (Sham Comparator): Sham stimulation - 10 sessions during 2 consecutive weeks
  Interventions: Device: Transorbital electrical stimulation (Eyetronic Next Wave 1.1) - Sham stimulation

INTERVENTIONS:
Device: Transorbital electrical stimulation (Eyetronic Next Wave 1.1) — Calibration phase: The patient will use a response button to indicate the threshold from which he feels a luminous sensation (phosphene). In a second step, he will use the same answer button to indicate the stimulation frequency from which the phosphenes become continuous.
  Stimulation phase: From these 2 parameters (amplitude and frequency), the stimulation session will begin for a duration of approximately 40 to 50 minutes, the settings being dependent of the individual thresholds.
  Arms: Active Transorbital electrical stimulation
Device: Transorbital electrical stimulation (Eyetronic Next Wave 1.1) - Sham stimulation — The calibration phase is identical to the active stimulation. During the stimulation phase, the operator will manually interrupt the stimulation 60 seconds after the start of the session.
  Arms: Sham Transorbital stimulation

SUMMARY:
In light of experimental models showing that neuronal electrical activity is crucial for the remyelination process, we hypothesize that maintenance of electrical axonal activity in the early stages of optic neuritis may promote myelin repair, limiting thereby axonal degeneration.

In humans, electrical stimulation of the optic nerve has been tested mainly in ischemic neuropathy and retinitis pigmentosa, which are both associated with severe axonal/retinal pathology and poor visual prognosis. In contrast, the inflammation of the optic nerve in optic neuritis is generally transient, with less severe axonal damage at the acute phase, which would allow for better efficacy of electrical stimulation as a strategy to promote remyelination and neuroprotection.In light of experimental models showing that neuronal electrical activity is crucial for the remyelination process, we hypothesize that maintenance of electrical axonal activity in the early stages of optic neuritis may promote myelin repair, limiting thereby axonal degeneration.

In humans, electrical stimulation of the optic nerve has been tested mainly in ischemic neuropathy and retinitis pigmentosa, which are both associated with severe axonal/retinal pathology and poor visual prognosis. In contrast, the inflammation of the optic nerve in optic neuritis is generally transient, with less severe axonal damage at the acute phase, which would allow for better efficacy of electrical stimulation as a strategy to promote remyelination and neuroprotection.

DETAILED DESCRIPTION:
This is a randomized, controlled, prospective, interventional, blinded trial which aims to evaluate the safety and efficacy of transorbital electrical nerve stimulation on remyelination and neuroprotection after an acute episode of retrobulbar optic neuritis in patients with multiple sclerosis (MS).

Expected Explorations: The study is composed of 14 visits: a screening/inclusion visit with neurological and ophthalmological evaluation, electrophysiology, MRI and Magnetoencephalography (MEG), 10 transorbital electrical stimulation or sham stimulation visits and finally 3 follow-up visits and evaluations (neurological and ophthalmological). Patient's participation will last 49 weeks (inclusion visit and 48 weeks of follow-up). Participation of healthy volunteers will last one day.

MS patients diagnosed with an optic neuritis will be randomized either in the active arm (transorbital electrical stimulation of the optic nerve - 10 sessions during 2 consecutive weeks) or in the placebo arm (sham stimulation - 10 sessions during 2 consecutive weeks) Expected benefits: Electrical stimulation of the optic nerve after an acute episode of retrobulbar optic neuritis may promote remyelination in the optic nerve and a better long-term visual outcome.

ELIGIBILITY:
Inclusion Criteria:

* For MS patients:
* Age between 18 and 60 years old.
* Relapsing Remitting MS (criteria of McDonald 2017) evolving for less than 10 years or Clinically Isolated Syndrome (CIS)-MS with criteria of spatial dissemination on MRI
* Subject presenting an acute unilateral episode of optic neuritis treated optimally (bolus of corticosteroids and plasma exchanges if considered necessary)
* Last medical treatment for optic neuritis received between 30 and 90 days before inclusion
* Visual acuity <7/10 of the affected eye at the time of inclusion
* Social security scheme or beneficiary of such a scheme

For Healthy Volunteers:

* Age between 18 and 60 years old.
* No history of neurological or ophthalmological diseases
* Corrected visual acuity ≥ 8/10
* Scheme or beneficiary of such a scheme

Exclusion Criteria:

For patients:

* Differential diagnosis of Optic neuritis:

  i) Atypical acute optic neuritis (papillitis, severe papilledema, initial optic atrophy) ii) Optic neuromyelitis iii) Normal VEP during the inclusion visit iv) No detection of VEP during the inclusion visit
* Impossibility to perform MRI, MEG, or electrical stimulation:

Pacemaker or neurosensory stimulator or implantable defibrillator Clip on an aneurysm or clip on a vascular malformation of the brain Cochlear implants Ocular or cerebral ferromagnetic foreign bodies Metal prostheses or metal clips or splinters Ventriculoperitoneal neurosurgical bypass valves Permanent makeup of the eyelids or lips Black tattoo, important and close to the cranio-facial sphere. Copper Intrauterine Device Person with proven claustrophobia Epilepsy Brain tumor Intraocular pressure without specific treatment Hypertension without treatment Acute retinal hemorrhage Periorbital skin irritation Significant cognitive deficit Known gadolinium allergy

* Person with severe or uncontrolled symptoms of kidney, liver, hematological, gastrointestinal, pulmonary or cardiac disease or any uncontrolled intercurrent disease at the time of inclusion.
* Pregnant or breath-feeding woman.
* Refusal of the participant to be informed in case of fortuitous discoveries having a direct impact on his health and requiring appropriate care
* person under judicial protection or deprived of liberty

For healthy volunteers:

* Contraindication to MRI or MEG
* Person with severe or uncontrolled symptoms of kidney, liver, hematological disease, gastrointestinal, pulmonary or cardiac disease or any uncontrolled intercurrent pathology at the time of inclusion.
* Pregnant or breath-feeding woman.
* Refusal of the participant to be informed in case of fortuitous discoveries having a direct impact on his health and requiring appropriate care
* Person under the protection of justice or deprived of liberty

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
P100 latency (VEP) after treatment | 24 weeks
  Modification of the latency of P100 wave measured by Visual Evoked Potential (VEP) after 24 weeks of treatment with electrical or sham stimulation.

SECONDARY OUTCOMES:
Change of P100 amplitude (VEP) after treatment | 24 weeks
  Modification of the amplitude of P100 wave measured by Visual Evoked Potential (VEP) after 24 weeks of treatment with electrical or sham stimulation.
Change of P100 latency and amplitude (VEP) after treatment | 12 and 48 weeks
  Modification of the latency and amplitude of P100 wave measured by Visual Evoked Potential (VEP) after 12 and 48 weeks of treatment with electrical or sham stimulation.
Evolution of macular volume after treatment | 12, 24 and 48 weeks
  Evolution since inclusion of macular volume (with Optical Coherence Tomography) at weeks 12, 24 and 48 after transorbital electrical treatment or sham stimulation.
Change of mean and temporal Retinal Nerve Fiber Layer (RNFL) thickness and average thickness of macular ganglion cell layer after treatment | 12, 24 and 48 weeks
  Evolution since inclusion of mean and temporal Retinal Nerve Fiber Layer (RNFL) thickness and average thickness of macular ganglion cell layer (with Optical Coherence Tomography) at weeks 12, 24 and 48 after transorbital electrical treatment or sham stimulation.
Change of average thickness of macular ganglion cell layer after treatment | 12, 24 and 48 weeks
  Evolution since inclusion of average thickness of macular ganglion cell layer (with Optical Coherence Tomography) at weeks 12, 24 and 48 after transorbital electrical treatment or sham stimulation.
Change of mean deflection of visual field 24-2 after treatment | 12, 24 and 48 weeks
  Change in the mean deflection of visual field 24-2 (24-2 Humphrey visual field analyser) at weeks 12, 24 and 48 compared to inclusion after electrical treatment or sham stimulation.
Occurrence of adverse events related or not to the stimulation | through study completion, an average of 3 years
  Reporting of adverse events related or not to the stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Céline Louapre, Principal Investigator — Institut du Cerveau et de la Moelle Epiniere, Pitie Salpetriere Hospital, Paris; Saddek Mohand-Said, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
Locations (2):
- France (2):
  - Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
  - Institut du Cerveau et de la Moelle epiniere - Hopital Pitie Salpetriere, Paris